CLINICAL TRIAL: NCT02834702
Title: Sinew Acupuncture for Chronic Mechanical Neck Pain: a Randomized Assessor-blind Sham-controlled Trial
Brief Title: Sinew Acupuncture for Neck Pain: Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHongKong-UW 15-456
Record Dates: First submitted 2016-07-13; First posted 2016-07-15 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Neck Pain
Keywords: sinew acupuncture; neck pain; chronic pain
MeSH Terms: conditions — Neck Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinew acupuncture (Experimental): Sinew acupuncture
  Interventions: Device: Sinew acupuncture
- Sham acupuncture (Sham Comparator): Sham acupuncture
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Sinew acupuncture — The subject is asked to be on sitting posture. The skin around the needling points is disinfected with a 75% alcohol swap. A tube-guided, sterilized, disposal needle is then inserted (at a small angle to the skin) into the acupoint at 0.5-1 cun (depending on point location and body size of the subject). No needle sensation (deqi sensation) is required. A piece of surgical adhesive tape will be applied to the needle immediately after insertion.
  Arms: Sinew acupuncture
Device: Sham acupuncture — The procedure in the sham acupuncture group will be as similar to that of the acupuncture group as possible. In the sham acupuncture group, however, a mock plastic needle guiding tube is tapped on the surface of each acupoint (Ashi point and traditional acupoints) to produce some discernible sensation. A piece of adhesive tape is immediately applied to fix the needle on the dermal surface tapped, without needle insertion. In addition, a plastic tube-guided needle is superficially inserted at the sham point at less than 5mm in depth.
  Arms: Sham acupuncture

SUMMARY:
The study aims to examine the efficacy and safety of sinew acupuncture for chronic mechanical neck pain (CMNP).

DETAILED DESCRIPTION:
Objectives:

Sinew acupuncture is a superficial needling technique with the advantage of minimal pain, feasible manipulation, and no apparent adverse effects. The proposal aims to examine the efficacy and safety of sinew acupuncture for chronic mechanical neck pain (CMNP).

Hypothesis to be tested:

Sinew acupuncture can reduce pain intensity, and improve neck pain disability and health-related quality of life without significant side effects for CMNP subjects compared to a sham acupuncture treatment.

Design:

A randomized, subject- and assessor-blind, sham acupuncture-controlled clinical trial

Participants:

Subjects (N=130) will be randomized into sinew acupuncture or sham acupuncture group (in 1:1 ratio).

Study instrument:

Visual Analog Scale (VAS), Northwick Park Neck Pain Questionnaire (NPQ) and Short Form-36 (SF-36)

Intervention:

Sinew acupuncture group will receive five sessions of needling in two weeks. Sham group will receive the non-invasive treatment with the same procedures. All subjects are followed up for 4 weeks.

Main outcome measures:

VAS for neck pain intensity at week 3 serves as the primary outcome. VAS at other time points, NPQ score and SF-36 at week 1, 2, 3, and 6, and adverse events are analyzed as the secondary outcomes.

Data analysis:

Analysis will be on the 'intention to treat' principle. T-test and mixed-effect model analysis will be used to measure primary and secondary outcomes respectively.

Expected results:

Five sessions of sinew acupuncture treatment can significantly reduce neck pain intensity, and improve neck pain disability and quality of life without obvious side effects.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18 years or above; (2) able to read and write Chinese; (3) the pain is located between the neck and shoulder regions and movement or palpation of the cervical region provokes the symptoms (18); (4) the pain has persisted for more than 3 months; (5) VAS (0 to 100 mm) pain score is ≥30 mm at baseline assessment; (6) no treatments (Chinese medicine, acupuncture, moxibustion, physiotherapies, medications, etc) intended for pain management have been received within the preceding two weeks.

Exclusion Criteria:

* (1) a history of fracture or surgery to the neck; (2) malignant tumor; (3) cervical congenital abnormality; (4) a severe psychiatric illness; (5) needle phobia; (6) acupuncture treatment in the preceding 3 months, and (7) other acupuncture contraindications as indicated in Hospital Authority Guideline on Safety in Acupuncture for Chinese Medicine Practitioners (Quality and Risk Sub-Committee, Hospital Authority, 2010).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | week 3
  VAS at week 3

SECONDARY OUTCOMES:
VAS | week 1, 2 & 6
  VAS at week 1, 2 & 6
Northwick Park Neck Pain Questionnaire (NPQ) | week 1, 2, 3 & 6
  NPQ at week 1, 2, 3 & 6
Short Form-36 (SF-36) | week 1, 2, 3 & 6
  SF-36 at week 1, 2, 3 & 6

OTHER OUTCOMES:
Adverse events | week 1, 2, 3 & 6
  Adverse events at week 1, 2, 3 & 6

CONTACTS AND LOCATIONS:
Overall Officials: Haiyong Chen, PhD, Principal Investigator — The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided